CLINICAL TRIAL: NCT02620449
Title: Impact of Lowering Phosphate Additive Intake on Metabolism and Cardiovascular Health in Community-Living Adults (Phosphate and Fibroblast Growth Factor 23 [FGF23]: Dietary and Molecular Mediators of Health and Disparities in Cardiovascular and Kidney Diseases)
Brief Title: Impact of Lowering Phosphate Additive Intake on Metabolism and Cardiovascular Health in Community-Living Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Orlando M. Gutierrez, MD, MMSc, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: F150728005
Record Dates: First submitted 2015-11-25; First posted 2015-12-03 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Healthy; Chronic Kidney Disease
Keywords: phosphorus; fibroblast growth factor 23; diet
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm study (Experimental)
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Participants will be fed a low-additive diet as the primary intervention

SUMMARY:
The purpose of the study is to learn more about how common food additives can affect phosphorus metabolism in people with normal kidney function and people with chronic kidney disease.

DETAILED DESCRIPTION:
Disturbances in phosphate homeostasis are strongly associated with cardiovascular morbidity and mortality. High dietary phosphate intake plays a central role in the development of disturbed phosphate metabolism and is common in persons consuming typical American diets rich in processed and fast foods. An important reason for the high phosphate content of these foods is the widespread use of phosphate-based food additives in the food supply. Phosphate additives are heavily utilized by the food manufacturing industry to enhance the appearance, taste and shelf-life of processed foods, accounting for as much as 50% of total phosphate intake per day. Prior work from our group suggest that high phosphate additive intake has serious cardiovascular consequences. We showed that phosphate excess induces heart disease and inflammation in experimental studies, and associates with heart disease and death independently of classic risk factors in epidemiology studies. Further, we showed that high phosphate additive intake stimulates the secretion of fibroblast growth factor 23 (FGF23), a phosphate-regulatory hormone directly implicated in the pathogenesis of cardiovascular disease. Together, these data strongly suggest that high phosphate additive intake promotes cardiovascular disease, with important potential implications for efforts to reduce disparities in cardiovascular disease. This is because individuals with low socioeconomic status have limited means to purchase healthy foods, resulting in excessive consumption of processed foods rich in phosphate additives. Moreover, low income neighborhoods have a disproportionately high prevalence of individuals with chronic kidney disease and black individuals, both groups that have impaired ability to excrete excess phosphate. Together, these data support our overriding hypothesis that high phosphate additive intake is a novel target for reducing socioeconomic and racial disparities in cardiovascular. We will test this hypothesis in detailed feeding studies of 80 individuals fed standardized meals with low phosphate additive content for 6 weeks. We will investigate the impact of reducing phosphate additive intake on changes in FGF23 levels, inflammatory markers and vascular function, and test for effect modification by race and chronic kidney disease (CKD). The results of these studies will help determine whether high phosphate additive intake is a modifiable risk factor for disparities in cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* (i.) Inclusion criteria for healthy volunteers: ≥18 years of age, normal kidney function (eGFR > 60 and normal urinalysis).

Exclusion Criteria:

* Exclusion criteria for healthy volunteers will include:

  * current smoking
  * extreme obesity (BMI ≥ 35 kg/m2)
  * pregnancy or breastfeeding
  * conditions affecting phosphate metabolism (e.g., hyper- or hypothyroidism; irregular menses for menstruating women)
  * current intake of medications that impact phosphate metabolism (high-dose vitamin D, chronic antacid use)
  * current use of blood pressure medications
  * abnormal serum phosphate (≥ 4.6 or < 2.5 mg/dl) or calcium levels (≥ 10.6 or < 8.5 mg/dl)
  * severe anemia (hemoglobin < 8 g/dl for women and < 9 g/dl for men).
  * Inability to receive weekly shipments of food at home.
  * Requirement for any special diet other than a regular diet.
  * Allergies to any foods in the standardized diets (ii.) Inclusion criteria for CKD patients: ≥18 years of age, eGFR 20-50 ml/min

Exclusion criteria for CKD patients will include:

* clinical need for a low potassium, low sodium or low protein diet
* new or recent change (<3 months) in dosage of medications known to impact vascular reactivity
* current smoking
* poorly controlled hypertension (≥160/100 mmHg)
* extreme obesity (BMI ≥ 35 kg/m2)
* pregnancy or breastfeeding
* conditions affecting phosphate metabolism (e.g., hyper- or hypothyroidism)
* current intake of medications that impact phosphate metabolism (e.g., high-dose vitamin D)
* abnormal serum phosphate (≥ 4.6 or < 2.5 mg/dl) or calcium levels (≥ 10.6 or < 8.5 mg/dl)
* severe anemia (hemoglobin < 8 g/dl for women and < 9 g/dl for men).
* Inability to receive weekly shipments of food at home.
* Allergies to any foods in the standardized diets

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08-28 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Change in circulating fibroblast growth factor 23 (FGF23) concentrations | 8 weeks
  Longitudinal change in FGF23 concentrations over 8 weeks
Change in brachial flow-mediated dilatation (FMD) | 8 weeks
  Longitudinal changes in FMD over 8 weeks
Change in pulse wave velocity (PWV) | 8 weeks
  longitudinal changes in PWV over 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Orlando Gutierrez, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Khan MB, Carnethon MR, Isakova T, Wolf M, Gutierrez OM. Effects of Lowering Dietary Phosphorus Additive Intake on Mineral Metabolism in Adults with and without CKD. Clin J Am Soc Nephrol. 2025 May 13;20(7):950-957. doi: 10.2215/CJN.0000000730. PMID 40359505